CLINICAL TRIAL: NCT02263885
Title: A Feasibility Clinical Trial of the Management of the Medically-Refractory Dyskinesia Symptoms of Advanced Idiopathic Parkinson's Disease With Unilateral Lesioning of the Globus Pallidum Using the ExAblate Transcranial System
Brief Title: ExAblate Transcranial MRgFUS of the Globus Pallidum for Treatment of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD002
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; ExAblate; MRgFUS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ExAblate Transcranial System (Experimental): Transcranial ExAblate MRgFUS
  Interventions: Device: ExAblate Transcranial System

INTERVENTIONS:
Device: ExAblate Transcranial System — Transcranial MRgFUS
  Other Names: MRgFUS; FUS; Focused Ultrasound; MR Guided Focused Ultrasound

SUMMARY:
The proposed study will evaluate the safety, and initial efficacy of using the ExAblate Transcranial to create a unilateral lesion in the globus pallidus as an adjunct to PD medications in subjects who are over 30 years of age and considered medication-refractory with advanced idiopathic Parkinson's disease (PD).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and initial clinical effectiveness of ExAblate Transcranial unilateral thermal ablation of the globus pallidus of subjects suffering from medication-refractory, advanced idiopathic PD.

Data will be collected to establish the basic safety and clinical efficacy of this type of treatment as the basis for later studies that will evaluate the full clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 30 years and older
* Subjects who are able and willing to give informed consent and able to attend all study visits through 24 Months
* Subjects with a diagnosis of idiopathic PD
* Levodopa responsive as defined by at least a 30% reduction in MDS-UPDRS motor subscale in the ON vs OFF medication state.
* Disabling motor complications of PD on optimum medical treatment
* Predominant disability from one side of the body (i.e unilateral or markedly asymmetric disease) as determined by movement disorders neurologist and neurosurgeon
* Subjects should be on a stable dose of all PD medications for 30 days prior to study entry.
* Subject is able to communicate sensations during the ExAblate Transcranial procedure.

Exclusion Criteria:

* Presence of other central neurodegenerative disease suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, corticobasal syndrome, dementia with Lewy bodies, and Alzheimer's disease.
* Any suspicion that Parkinsonian symptoms are a side effect from neuroleptic medications.
* Subjects who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia
* Unstable psychiatric disease, defined as active uncontrolled depressive symptoms, psychosis, delusions, hallucinations, or suicidal ideation. Subjects with stable, chronic anxiety or depressive disorders may be included provided their medications have been stable for at least 60 days prior to study entry and if deemed appropriately managed by the site neuropsychologist
* Subjects with significant depression as determined following a comprehensive assessment by a neuropsychologist.
* Legal incapacity or limited legal capacity as determined by the neuropsychologist
* Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse
* Subjects with unstable cardiac status including:

  1. Unstable angina pectoris on medication
  2. Subjects with documented myocardial infarction within six months of protocol entry
  3. Significant congestive heart failure defined with ejection fraction < 40
  4. Subjects with unstable ventricular arrhythmias
  5. Subjects with atrial arrhythmias that are not rate-controlled
* Severe hypertension (diastolic BP > 100 on medication)
* Current medical condition resulting in abnormal bleeding and/or coagulopathy
* Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
* Subjects with risk factors for intraoperative or postoperative bleeding as indicated by: platelet count less than 100,000 per cubic millimeter, a documented clinical coagulopathy, or INR coagulation studies exceeding the institution's laboratory standard
* Patient with severely impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2 (or per local standards should that be more restrictive) and/or who is on dialysis;
* Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Significant claustrophobia that cannot be managed with mild medication.
* Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment.
* History of intracranial hemorrhage
* History of multiple strokes, or a stroke within past 6 months
* Subjects with a history of seizures within the past year
* Subjects with brain tumors
* Subjects with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment.
* Are participating or have participated in another clinical trial in the last 30 days
* Any illness that in the investigator's opinion preclude participation in this study.
* Subjects unable to communicate with the investigator and staff.
* Pregnancy or lactation.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2019-05-15 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford University Medical Center, Stanford, California
  - University of Maryland Medical System, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - The Ohio State Wexner Medical Center, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Eisenberg HM, Krishna V, Elias WJ, Cosgrove GR, Gandhi D, Aldrich CE, Fishman PS. MR-guided focused ultrasound pallidotomy for Parkinson's disease: safety and feasibility. J Neurosurg. 2020 Nov 27;135(3):792-798. doi: 10.3171/2020.6.JNS192773. Print 2021 Sep 1. PMID 33481557

RESULTS

PARTICIPANT FLOW:
Groups:
- ExAblate Transcranial System Test Arm: Transcranial ExAblate MRgFUS
  Transcranial MRgFUS lesioning of the Globus Pallidum
Period: Overall Study
Arm/Group | ExAblate Transcranial System Test Arm
Started | 20
Completed | 10
Not Completed | 10
Not completed — Withdrawal by Subject | 7
Not completed — Alternative Treatment | 3

BASELINE CHARACTERISTICS:
Arm/Group | ExAblate Transcranial System Test Arm
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 18
  Race: Black | 0
  Race: Hispanic | 2
  Race: Other | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: The primary outcome of this feasibility trial was safety. Adverse Events were categorized by physicians as mild, moderate, or severe. Events resulting in impairment, requiring intervention to preclude impairment, or that were life threatening, and deaths were reported by physicians as Serious Adverse Events. Outcomes are entered in the adverse events module.
Time Frame: Month 24
Measure: Number; unit: Number of Adverse Events
Arm/Group | ExAblate Transcranial System Test Arm
Number analyzed (Participants) | 20
Number of Adverse Events | 36

2. Secondary Outcome: Unified Dyskinesia Rating Scale Total Score.
Description: The Unified Dyskinesia Rating Scale Total score assesses overall involuntary movements associated with the treatment of Parkinson's disease. The minimum score possible is 0. The maximum total score possible is 104. High scores show worse symptoms.
Time Frame: Screening, Month 3, Month 6, Month 12, Month 24
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ExAblate Transcranial System
Number analyzed (Participants) | 20
score on a scale
  Screening | 36.1 [31.2 to 40.9]
  Month 3 | 14.9 [9.3 to 20.4]
  Month 6 | 16.9 [10.1 to 23.7]
  Month 12 | 19.5 [11.9 to 27.1]
  Month 24 | 23.1 [12.4 to 33.8]

3. Secondary Outcome: Unified Dyskinesia Rating Scale (UDysRS), Part III
Description: The Unified Dyskinesia Ratient Scale (UDysRS) was developed to assess involuntary movements often associated with the treatment of Parkinson's disease. Part III evaluates the intensity of impairment of dyskinesia with respect to the performance of 7 tasks on a scale of 0 to 4. The sum of the Part III score ranges 0 to 28 and high scores show worse symptoms.
Time Frame: Screening, Month 3, Month 6, Month 12, Month 24
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ExAblate Transcranial System Test Arm
Number analyzed (Participants) | 20
score on a scale
  Screening | 10.2 [7.5 to 12.9]
  Month 3 | 4.5 [2.4 to 6.6]
  Month 6 | 6.0 [2.7 to 9.4]
  Month 12 | 4.1 [1.7 to 6.7]
  Month 24 | 5.8 [2.3 to 9.2]

4. Secondary Outcome: Movement Disorders Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part III Motor Exam
Description: The Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS UPDRSP Part III motor exam focuses specifically on the treated side tremor and motor fluctuations. Each of 11 items are scored from 0 to 4 for a total score minimum of 0 and a maximum of 44 points. High scores show worse symptoms.
Time Frame: Screening, Month 3, Month 6, Month 12, Month 24
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ExAblate Transcranial System Test Arm
Number analyzed (Participants) | 20
score on a scale
  Screening | 20.0 [17.5 to 22.4]
  Month 3 | 10.6 [8.7 to 12.5]
  Month 6 | 11.1 [9.6 to 12.6]
  Month 12 | 10.5 [8.2 to 12.7]
  Month 24 | 12.3 [9.8 to 14.9]

5. Secondary Outcome: Mood Disorders Society - Unified Parkinson's Disease Rating Scale Part II
Description: .Part II of the Mood Disorders Society Unified Parkinson's Disease Rating Scale focuses on the impact of symptoms on motor aspects of daily living. Part II consists of 13 items scored from 0 to 4 for a maximum score of 52. High Part II scores indicate worse (greater) impact.
Time Frame: Screening, Month 3, Month 6, Month 12, Month 24
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ExAblate Transcranial System Test Arm
Number analyzed (Participants) | 20
score on a scale
  Screening | 14.0 [10.7 to 17.3]
  Month 3 | 7.4 [5.14 to 9.6]
  Month 6 | 8.7 [5.1 to 10.8]
  Month 12 | 11.4 [8.6 to 14.2]
  Month 24 | 13.8 [9.4 to 18.2]

6. Secondary Outcome: Mood Disorder Society Unified Parkinson's Disease Rating Scale Part IV
Description: Part IV of the Mood Disorder Society Unified Parkinson's Disease Rating Scale assesses dyskinesias that include OFF-state dystonia; items include time spent with dyskinesia, functional impact of dyskinesia, time spent in the OFF state, functional impact of fluctuations, complexity of motor fluctuations and painful OFF state dystonia. Six items are scored 0 to 4 with a maximum total score of 24. High scores indicate worse symptoms.
Time Frame: Screening, Month 3, Month 6, Month 12, Month 24
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ExAblate Transcranial System Test Arm
Number analyzed (Participants) | 20
score on a scale
  Screening | 11.1 [8.6 to 13.6]
  Month 3 | 6.4 [4.5 to 8.2]
  Month 6 | 6.0 [4.4 to 7.6]
  Month 12 | 5.9 [4.0 to 7.8]
  Month 24 | 8.7 [5.8 to 11.5]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 24 months.
Arm/Group | ExAblate Transcranial System Test Arm
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate Transcranial System Test Arm (N=20)
Stroke (Nervous system disorders) | 1 (1) — A subject experienced a stroke 2 years post-treatment. The DSMB adjudicated the stroke as unrelated to the device or procedure.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate Transcranial System Test Arm (N=20)
Bruise (Skin and subcutaneous tissue disorders) | 2 (2) — Bruise unrelated to device or procedure
Facial Edema (Skin and subcutaneous tissue disorders) | 3 (3) — Edema related to stereotactic frame
Drooling (General disorders) | 2 (2) — Drooling related to Parkinson's Disease
Dyskinesia (Nervous system disorders) | 2 (2) — Dyskinesia related to Parkinson's Disease
Nausea/Vomiting (Gastrointestinal disorders) | 3 (3) — Tranient nausea/vomiting, resolving within 72 hours of treatment
Headache (General disorders) | 3 (3) — Transient headache, resolving within 72 hours of treatment
Sonication Related Head Pain (General disorders) | 7 (7) — Transient sonication related head pain, resolving within 72 hours of treatment.
Fine Motor Problems (Nervous system disorders) | 2 (2)
Headache (General disorders) | 5 (5) — Procedure related headache
Anxiety (Psychiatric disorders) | 2 (2) — Procedure related anxiety
Dysarthria (Nervous system disorders) | 4 (4) — Pallidotomy related dysarthria

LIMITATIONS AND CAVEATS:
This is a single-arm, open label, feasibility trial. Analyses included basic descriptive statistics. No hypothesis testing was proposed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/85/NCT02263885/Prot_SAP_000.pdf